CLINICAL TRIAL: NCT05933603
Title: Medications for Obstructive Sleep Apnea to Improve Cognition in Children With Down Syndrome
Acronym: MOSAIC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1908864846v2; R33HL151254 (NIH)
Record Dates: First submitted 2023-06-26; First posted 2023-07-06 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Obstructive Sleep Apnea; Down Syndrome
MeSH Terms: conditions — Sleep Apnea, Obstructive; Down Syndrome | interventions — Atomoxetine Hydrochloride; oxybutynin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ato-oxy (Experimental): 0.5 mg/kg (max 40 mg) atomoxetine and 5 mg oxybutynin
  Interventions: Drug: Atomoxetine and Oxybutynin (ato-oxy)

INTERVENTIONS:
Drug: Atomoxetine and Oxybutynin (ato-oxy) — 0.5 mg/kg atomoxetine (max 40 mg) and 5 mg oxybutynin by mouth nightly

SUMMARY:
This is an open-label study of the combination of atomoxetine and oxybutynin (ato-oxy) in children with Down syndrome and obstructive sleep apnea (OSA) documented by polysomnography (PSG). Participants will receive ato-oxy for 6 months. Ato-oxy dose will be 5 mg oxybutynin and 0.5mg/kg/day (max 40 mg) atomoxetine. Dosing of the study treatment will occur approximately 30 minutes prior to bedtime. Participants who withdraw from the study will not be replaced.

Study participants will undergo eligibility screening that will include an initial screening to determine whether non- PSG enrollment criteria are met, followed by a 1 night in-lab PSG and health-related quality of life (HRQOL) and cognitive assessment for participants who qualify based on non-PSG criteria. For participants who are eligible and enroll in the study, the screening PSG night will serve as the baseline measure for apnea hypopnea index (AHI) and other PSG endpoints. On the final night of dosing for ato-oxy participants will return for inpatient PSG and health-related quality of life assessment and cognitive assessment. The primary efficacy endpoint is the change in obstructive AHI from baseline.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants between 6 to 17 years of age, inclusive, at the Screening Visit.
2. Known diagnosis of Down syndrome (trisomy 21, but not translocation or mosaicism)

Exclusion Criteria:

1. Presence of central sleep apnea on polysomnography (central AHI ≥ 5)
2. Currently using and adherent to positive airway pressure therapy (>4 hours per night for 70% of nights in the past 30 days based on device download or parent report)
3. Monoamine oxidase inhibitor use
4. Urinary retention
5. Prematurity < 32 weeks estimated gestational age
6. Seizure disorder
7. Untreated or inadequately treated hypothyroidism
8. Significant traumatic brain injury
9. Congenital heart disease and not cleared to participate by the patient's cardiologist
10. History of current, untreated depression
11. History of liver disease
12. 3+ or greater tonsillar hypertrophy
13. Positive urine pregnancy test
14. Hypoxemia independent of respiratory events on baseline polysomnography (≥5 minutes with oxygen saturation <90%)
15. Presence of central sleep apnea on baseline polysomnography (central AHI ≥ 5)

3. Absence of OSA defined as total AHI <5 on baseline polysomnography

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Estimated)
Dates: Start 2023-09-29 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
obstructive apnea-hypopnea index (oAHI) | 6 months
  change in number of obstructive apneas and hypopneas per hour on polysomnography from baseline (% change)

SECONDARY OUTCOMES:
Obstructive Sleep Apnea-18 score (OSA-18) | 6 months
  Change in OSA-18 (a measure of health-related quality of life) from baseline. The OSA-18 score ranges from 18 to 136, with lower scores indicating better health-related quality of life.
Paired Associates Learning test | 6 months
  Change in Paired Associate Learning test total errors (a measure of memory) from baseline

OTHER OUTCOMES:
Pediatric Quality of Life Inventory (PedsQL) total score | 6 months
  Change in PedsQL total score (a measure of health-related quality of life) from baseline. The PedsQL score ranges from 0-100, with higher scores indicating better health-related quality of life.
Processing speed | 6 months
  Change in processing speed as measured by A-MAP from baseline
Verbal IQ | 6 months
  Change in verbal IQ as measured by the Kaufman Brief IQ Test 2 from baseline
Verbal memory | 6 months
  Change in verbal memory as measured by A-MAP from baseline
Language | 6 months
  Change in child vocalizations/ hour as measured by LENA
Caregiver Global Impression of Change | 6 months
  Change in Caregiver Global Impression of Change from baseline. This will be assessed on a seven point scale answering the question: Since the start of this therapy, my child's overall status is: 1. Very much improved; 2. Much improved; 3. Minimally Improved; 4. No change; 5. Minimally worse; 6. Much worse or 7. Very much worse.
N1 sleep percentage | 6 months
  Change in N1 sleep percentage on polysomnography from baseline
REM sleep percentage | 6 months
  Change in REM sleep percentage on polysomnography from baseline
N3 sleep percentage | 6 months
  Change in N3 sleep percentage on polysomnography from baseline
Arousal Index | 6 months
  change in number of arousals per hour on polysomnography from baseline
Executive Function | 6 months
  Change in Behavior Rating Inventory of Executive Function (BRIEF) Global Executive Composite from baseline
Adaptive function | 6 months
  Change in Vineland 3 adaptive behavior composite scale from baseline
Attention Deficit Hyperactivity Disorder symptoms | 6 months
  Change in Conners-3 Attention Deficit Hyperactivity Disorder Index from baseline

CONTACTS AND LOCATIONS:
Locations (1):
- University of Arizona, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be made available via a database such as sleepdata.org.
Time Frame: Data will be made available following primary analysis and publication of primary study results.